CLINICAL TRIAL: NCT04907539
Title: A Multi-arm, Phase II, Open-Label, Multicentre Study to Assess the Preliminary Efficacy of RXC004 in Monotherapy and in Combination With Nivolumab, in Patients With Ring Finger Protein 43 (RNF43) or R-spondin (RSPO) Aberrated, Metastatic, Microsatellite Stable, Colorectal Cancer Who Have Progressed Following Therapy With Current Standard of Care (PORCUPINE)
Brief Title: A Study to Assess Efficacy of RXC004 +/- Nivolumab in Ring Finger Protein 43 (RNF43) or R-spondin (RSPO) Aberrated, Metastatic, Microsatellite Stable, Colorectal Cancer After Progression on Standard of Care (SOC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Redx Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RXC004/0002
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
Keywords: Open label; RXC004; Nivolumab; Ring finger protein 43; R-spondin; Efficacy; Safety; Pharmacokinetics
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: RXC004 monotherapy (Experimental): Patients will receive RXC004 (2 mg once daily [QD], orally).
  Patients in Arm A may crossover to Arm B treatment if they have progressive disease on the first Response Evaluation Criteria in Solid Tumours, (RECIST) scan (if Arm B is open at the time of progression).
  Interventions: Drug: RXC004; Biological: Denosumab
- Arm B: RXC004 + nivolumab (Experimental): Patients will receive RXC004 (1.5 mg QD, orally) in combination with nivolumab (480 mg every 4 weeks [q4w], intravenous [IV] infusion).
  Arm B will be opened once a RP2D for RXC004 in combination with nivolumab is established in the phase I dose escalation study (NCT03447470). RXC004 dose to be used in combination with nivolumab will be based on data from the phase 1 study (NCT03447470).
  Interventions: Drug: RXC004; Biological: Nivolumab; Biological: Denosumab

INTERVENTIONS:
Drug: RXC004 — RXC004 will be administered orally, 2 mg QD (Monotherapy); and 1.5 mg QD (Combination therapy)
  Dose Formulation: 0.5 mg or 1 mg capsules.
Biological: Nivolumab — Nivolumab will be administered via IV infusion, 480 mg q4w.
  Arms: Arm B: RXC004 + nivolumab
Biological: Denosumab — Denosumab will be administered via subcutaneous (SC) injection, 120 mg once every month.
  Use: Prophylactic

SUMMARY:
This is a Phase II, open label, multicentre, multi-arm, study to evaluate the preliminary efficacy and safety of RXC004 as monotherapy and in combination with nivolumab in patients with Ring finger protein 43 (RNF43) or R-spondin (RSPO) aberrated, microsatellite stable (MSS), colorectal cancer (CRC), that have progressed following current standard of care treatment.

DETAILED DESCRIPTION:
The study is composed of two arms, RXC004 monotherapy (Arm A) and RXC004 in combination with nivolumab (Arm B). 20 evaluable patients will be enrolled in Arm A and 20 eligible patients in Arm B.

The study initially opened with Arm A; Arm B will be opened once a recommended Phase II dose (RP2D) for RXC004 in combination with nivolumab is established in the phase I dose escalation study (NCT03447470).

Once Arm B is opened, patients who are eligible for both Arm A and Arm B will be randomised 2:1 to Arm B: Arm A in an open-label manner.

Patients in Arm A may be treated with RXC004 + nivolumab if they have progressive disease on the 8 week scan, as long as they are eligible for Arm B and have Sponsor approval.

ELIGIBILITY:
Inclusion Criteria:

* Histological documentation of metastatic (Stage IV) Colorectal cancer (CRC) and

  1. Documented tumour tissue aberration in RNF43 and/or RSPO
  2. Documented confirmation of microsatellite stable (MSS) status
* Patients must have had documented radiological progression following a minimum of 1 prior SOC treatment regimen for metastatic disease
* Eastern Cooperative Oncology Group performance status 0 or 1
* At least one lesion that is measurable by RECIST 1.1 at baseline
* Patients must have at least one lesion suitable for biopsy at screening and be willing to provide mandatory tumour biopsy samples
* Patients with adequate organ functions
* Female patients of childbearing potential must have a negative pregnancy test prior to start of dosing
* Female patients of childbearing potential and male patients with female partners of childbearing potential must agree to use a highly effective method of contraception during the study and for at least 5 months after the last dose of study drug.

For patients on RXC004 monotherapy treatment (Arm A) the following inclusion criteria will also apply to enter the RXC004 + nivolumab treatment phase:

* Patients must have had documented RECIST1.1 defined radiological progression on RXC004 monotherapy treatment on the first scheduled scan (week 8 +/- 1 week)
* Patients must receive Cycle 1 Day 1 of combination study treatment within 28 days of the first scheduled scan (week 8 +/- 1 week).

Exclusion Criteria:

* Prior therapy with a compound of the same mechanism of action as RXC004
* Patients at higher risk of bone fractures
* Any known uncontrolled inter-current illness or persistent clinically significant toxicity related to prior anti-cancer treatment
* Patients who have any history of an active (requiring treatment) other malignancy within 2 years of study entry
* Patients with known or suspected brain metastases
* Use of anti-neoplastic agents, immunosuppressants and other investigational drugs
* Patients with a known hypersensitivity to any RXC004 excipients
* Patients with a contra-indication for denosumab treatment
* Patients who are pregnant or breast-feeding
* Use of any live or live-attenuated vaccines against infectious diseases (e.g., influenza nasal spray, varicella) within 4 weeks (28 days) of initiation of study treatment
* Patients with a mean resting corrected QTcF >470 ms, obtained from triplicate electrocardiograms performed at screening

For patients on RXC004 + nivolumab combination treatment (Arm B or Arm A RXC004 + nivolumab treatment phase):

* Patients with any contraindication to the use of nivolumab
* Patients with active or prior documented autoimmune or inflammatory disorders within the past 5 years
* Patients with active infections, including tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus
* Patients with a history of allogeneic organ transplant or active primary immunodeficiency
* Patients with a known hypersensitivity to nivolumab or any of the excipients of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (5):
  - Providence Medical Foundation, Santa Rosa, California
  - Community Health Network Cancer Center North - Community Hospital Network, Indianapolis, Indiana
  - OptumCare Cancer Care, Las Vegas, Nevada
  - UT MD Anderson Cancer Center, Houston, Texas
  - Lumi Research, Kingswood, Texas
- South Korea (5):
  - National Cancer Center, Goyang-si, Gyeonggido [Kyonggi-do]
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System - Medical Oncology, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Samsung Medical Center - Hematology-Oncology, Seoul
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Clìnic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (7):
  - Beatson West of Scotland Cancer Centre - Oncology, Glasgow, Scotland
  - Queen Elizabeth Hospital - Clinical Reasearch, Birmingham
  - University College of London (UCL), London
  - The Royal Marsden NHS Foundation Trust - Royal Marsden Hospital, London
  - Christie Hospital, Manchester
  - Oxford Cancer Centre, Oxford
  - The Royal Marsden Hospital (Surrey), Surrey Quays

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 08 November 2021 to 02 April 2024 at multiple centers in 4 countries (South Korea, Spain, United Kingdom and United States of America).
Pre-assignment Details: Patients who met the inclusion criteria, and none of the exclusion criteria were enrolled to the study. All study assessments were performed as per the Schedule of Assessment.
Groups:
- Arm A: RXC004 Monotherapy: Patients received 2 mg of RXC004 monotherapy once daily orally.
- Arm B: RXC004+Nivolumab: Patients received 1.5 mg of RXC004 once daily along with the combination of 480 mg of Nivolumab every 4 weeks orally.
Period: Overall Study
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Started | 17 | 8
Completed | 2 | 5
Not Completed | 15 | 3
Not completed — Consent withdrawn | 1 | 0
Not completed — Death | 14 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab | Total
Number analyzed (Participants) | 17 | 8 | 25
Age, Continuous [Mean (Standard Deviation); unit: Year] | 53.4 (13.87) | 64.8 (7.78) | 57.0 (13.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 9 | 3 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — For a single patient of a particular ethnicity, the data was not reported under specific ethnicity in specific arm, rather customized option was used, and the data was reported as "Other" to maintain patient's confidentiality
  Participants
    Not Hispanic or Latino | 14 | 6 | 20
    Not Stated | 1 | 1 | 2
    Unknown | 1 | 0 | 1
    Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: RXC004 Monotherapy (Arm A): Disease Control Rate (DCR) Using Each Patient's Best Overall Response (BOR) According to Response Evaluation Criteria in Solid Tumours, Version 1.1 (RECIST 1.1)
Description: The anti-tumour activity of RXC004 monotherapy was evaluated. DCR is defined as the percentage of patients with a BOR of either complete response (CR), partial response (PR) or stable disease (SD) for at least 16 weeks post baseline.
Time Frame: Up to 28 months
Population: Evaluable set consisted of all patients who received radiographic assessment at baseline (with measurable disease according to RECIST 1.1), received at least 4 weeks of study treatment and at least 1 post-dose radiographic tumour assessment or progressed or died ahead of the first radiographic assessment. Patients with important protocol deviations that may have impacted outcome were excluded from the population.
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm A: RXC004 Monotherapy
Number analyzed (Participants) | 11
Percentage of patients | 18.2 [3.33 to 47.01]

2. Primary Outcome: RXC004+Nivolumab Combination Therapy (Arm B): Objective Response Rate (ORR) Using Each Patient's BOR According to RECIST 1.1
Description: The anti-tumour activity as a combination therapy of RXC004 +nivolumab was evaluated. ORR is defined as the percentage of patients with a BOR of CR or PR based on local investigator assessment, as defined in RECIST 1.1.
Time Frame: Up to 28 months
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 7
Percentage of patients | 14.3 [0.73 to 52.07]

3. Secondary Outcome: Best Percentage Change in Tumor Size
Description: The preliminary efficacy of RXC004 monotherapy and combination therapy of RXC004 + nivolumab was evaluated. The best percentage change in tumour size was determined at a patient level. Percentage change in tumour size was derived at each visit by the percentage change from baseline in the sum of diameters of target lesions. The best percentage change in tumour size was the patients value representing the largest decrease (or smallest increase) from baseline in tumour size.
Time Frame: Up to 28 months
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage change in tumor size
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 11 | 7
Percentage change in tumor size | 9.34 [-11.8 to 59.8] | 0.00 [-40.4 to 39.4]

4. Secondary Outcome: Progression Free Survival (PFS)
Description: The preliminary efficacy of RXC004 monotherapy and combination therapy of RXC004 + nivolumab was evaluated. PFS is defined as the time from first dose of study treatment until the date of disease progression or death (by any cause in the absence of progression).
Time Frame: Up to 28 months
Population: Full analysis set consisted of all patients who were enrolled and received at least one dose of study drug (RXC004).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 17 | 8
Months | 2.0 [1.31 to 2.33] | 3.9 [1.58 to NA] — Due to insufficient number of patients with events, estimates were not calculable using methodology specified in Statistical Analysis Plan (SAP).

5. Secondary Outcome: Duration of Response (DOR)
Description: The preliminary efficacy of RXC004 monotherapy and combination therapy of RXC004 + nivolumab was evaluated. The DOR is as the time from the date of first documented response until date of documented progression or death in the absence of disease progression. DOR was not calculated as 1 patient had PR, and 0 patient had CR. As pre-specified in the SAP that after the review of the available data, DOR would not be summarized and listed.
Time Frame: Up to 28 months
Population: Evaluable set consisted of all patients who received radiographic assessment at baseline (with measurable disease according to RECIST 1.1) received at least 4 weeks of treatment and at least 1 post-dose radiographic tumour assessment or progressed or died ahead of the first radiographic assessment. Patients with important protocol deviations that may impact outcome were excluded from population.
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: RXC004 Monotherapy (Arm A): Objective Response Rate (ORR) Using Investigator Assessments According to RECIST 1.1
Description: The preliminary efficacy of RXC004 monotherapy was evaluated. ORR is defined as the percentage of patients with a BOR of CR or PR based on local investigator assessment as defined in RECIST 1.1.
Time Frame: Up to 28 months
Population: Evaluable set consisted of all patients who received radiographic assessment at baseline (with measurable disease according to RECIST 1.1), received at least 4 weeks of study treatment and at least 1 post-dose radiographic tumour assessment or progressed or died ahead of the first radiographic assessment. Patients with important protocol deviations that may impact outcome were excluded from the population.
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm A: RXC004 Monotherapy
Number analyzed (Participants) | 11
Percentage of patients | 0 [0.00 to 23.84]

7. Secondary Outcome: RXC004 + Nivolumab Combination Therapy (Arm B): Disease Control Rate Using Investigator Assessments According to RECIST 1.1
Description: The preliminary efficacy of combination therapy of RXC004 + nivolumab was evaluated. DCR is defined as the percentage of patients with a BOR of either CR, PR or SD for at least 16 weeks post baseline.
Time Frame: Up to 28 months
Population: as for outcome 6
Measure: Number (90% Confidence Interval); unit: Percentage of patients
Arm/Group | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 7
Percentage of patients | 57.1 [22.53 to 87.12]

8. Secondary Outcome: Overall Survival (OS)
Description: The preliminary efficacy of RXC004 monotherapy and combination therapy of RXC004 + nivolumab was evaluated. OS is defined as the time from first day of study treatment until death due to any cause.
Time Frame: Up to 28 months
Population: Full analysis set consisted of all patients who were enrolled and received at least one dose of study drug (RXC004).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 17 | 8
Months | 4.8 [1.3 to 6.5] | NA [1.7 to NA] — Due to insufficient follow-up information, the median for Arm B was not reached and the estimates were not calculable as per methodology specified in SAP.

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The pharmacokinetic (PK) (Cmax) of RXC004 in monotherapy and in combination therapy with nivolumab was evaluated.
Time Frame: On Cycle 0 Day 1 (3-7 days cycle in length) and Cycle 1 Day 15 (28 days cycle in length)
Population: The PK Analysis Set included all patients in the full analysis set with at least 1 blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 17 | 8
nanogram per milliliter (ng/mL)
  Cycle 0 Day 1: number analyzed (Participants) | 16 | 8
  Cycle 0 Day 1 | 65.2 (62.0) | 56.5 (56.4)
  Cycle 1 Day 15: number analyzed (Participants) | 11 | 7
  Cycle 1 Day 15 | 80.0 (66.8) | 79.4 (42.7)

10. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: The PK (Tmax) of RXC004 in monotherapy and in combination therapy with nivolumab was evaluated.
Time Frame: On Cycle 0 Day 1 (3-7 days cycle in length) and Cycle 1 Day 15 (28 days cycle in length)
Population: The PK Analysis Set included all patients in the full analysis set with at least 1 blood sample.
Measure: Median (Full Range); unit: Hour (h)
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 17 | 8
Hour (h)
  Cycle 0 Day 1: number analyzed (Participants) | 16 | 8
  Cycle 0 Day 1 | 2.07 [0.983 to 4.18] | 1.95 [0.933 to 2.12]
  Cycle 1 Day 15: number analyzed (Participants) | 11 | 7
  Cycle 1 Day 15 | 1.35 [0.517 to 6.12] | 1.98 [1.02 to 10.4]

11. Secondary Outcome: Minimum Observed Concentration Across the Dosing Interval (Cmin)
Description: The PK (Cmin) of RXC004 in monotherapy and in combination therapy with nivolumab was evaluated.
Time Frame: On Cycle 1 Day 15 (28 days cycle in length)
Population: The PK Analysis Set included all patients in the full analysis set with at least 1 blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 11 | 7
ng/mL | 12.8 (65.8) | 17.2 (49.4)

12. Secondary Outcome: Terminal Rate Constant (λz)
Description: The PK (λz) of RXC004 in monotherapy and in combination therapy with nivolumab was evaluated.
Time Frame: On Cycle 0 Day 1 (3-7 days cycle in length)
Population: The PK Analysis Set included all patients in the full analysis set with at least 1 blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hour
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 11 | 8
1/hour | 0.0769 (73.3) | 0.0540 (29.8)

13. Secondary Outcome: Terminal Half-life (t½)
Description: The PK (t½) of RXC004 in monotherapy and in combination therapy with nivolumab was evaluated.
Time Frame: On Cycle 0 Day 1 (3-7 days cycle in length)
Population: The PK Analysis Set included all patients in the full analysis set with at least 1 blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 11 | 7
hour (h) | 9.02 (73.3) | 12.2 (27.7)

14. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero to Infinity (AUC0-∞)
Description: The PK (AUC0-∞) of RXC004 in monotherapy and in combination therapy with nivolumab was evaluated.
Time Frame: On Cycle 0 Day 1 (3-7 days cycle in length)
Population: The PK Analysis Set included all patients in the full analysis set with at least 1 blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (h*ng/mL)
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 10 | 6
hour*nanogram/milliliter (h*ng/mL) | 733 (48.9) | 749 (45.0)

15. Secondary Outcome: Total Plasma Clearance After Oral Administration (CL/F)
Description: The PK (CL/F) of RXC004 in monotherapy and in combination therapy with nivolumab was evaluated.
Time Frame: On Cycle 0 Day 1 (3-7 days cycle in length)
Population: The PK Analysis Set included all patients in the full analysis set with at least 1 blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour (mL/h)
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 10 | 6
milliliter per hour (mL/h) | 2730 (48.9) | 2000 (45.0)

16. Secondary Outcome: Apparent Volume of Distribution After Oral Administration (Vz/F)
Description: The PK (Vz/F) of RXC004 in monotherapy and in combination therapy with nivolumab was evaluated.
Time Frame: On Cycle 0 Day 1 (3-7 days cycle in length)
Population: The PK Analysis Set included all patients in the full analysis set with at least 1 blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter (mL)
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 10 | 6
milliliter (mL) | 32300 (89.6) | 35800 (22.0)

17. Secondary Outcome: Number of Patients With Adverse Events (AEs)
Description: The safety and tolerability profile of RXC004 monotherapy and RXC004 + nivolumab combination was evaluated. The grading scales found in the revised National Cancer Institute Common Terminology Criteria for Adverse events (CTCAE) latest version was utilized for all events with an assigned CTCAE grading. Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL; Grade 4: Life-threatening, urgent intervention required; Grade 5: Death related to AE.
Time Frame: From time of signature of informed consent form throughout the treatment period and until 30 days after the last dose of RXC004 (for RXC004 monotherapy only) or 90 days after the last dose of Nivolumab (for RXC004 + nivolumab) (up to 28 months)
Population: The safety analysis set consisted of all patients who were enrolled and received at least one dose of study drug (RXC004).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
Number analyzed (Participants) | 17 | 8
Participants
  Treatment emergent adverse event (TEAE) | 17 | 8
  RXC004 Related TEAE | 14 | 8
  Nivolumab Related TEAE | 1 | 5
  Grade >=3 TEAE | 9 | 5
  RXC004 Related Grade >=3 TEAE | 3 | 4
  Nivolumab Related Grade >=3 TEAE | 0 | 2
  Serious TEAE | 3 | 5
  RXC004 Related Serious TEAE | 2 | 4
  Nivolumab Related Serious TEAE | 0 | 2
  TEAE Leading to Death | 0 | 1
  TEAE Leading to Permanent Discontinuation or Reduction or Interruption of RXC004 | 10 | 7
  TEAE Leading to Permanent Discontinuation of RXC004 | 2 | 3
  TEAE Leading to Reduction of RXC004 | 3 | 4
  TEAE Leading to Interruption of RXC004 | 8 | 3
  TEAE Leading to Permanent Discontinuation or Interruption of Nivolumab | 0 | 5
  TEAE Leading to Permanent Discontinuation of Nivolumab | 0 | 3
  TEAE Leading to Interruption of Nivolumab | 0 | 3

ADVERSE EVENTS:
Time Frame: From time of signature of informed consent form throughout the treatment period and until 30 days after the last dose of RXC004 (for RXC004 monotherapy only) or 90 days after the last dose of Nivolumab (for RXC004 + nivolumab) (up to 28 months)
Description: Safety Set included all patients who were enrolled and received at least one dose of study drug (RXC004).
Arm/Group | Arm A: RXC004 Monotherapy | Arm B: RXC004+Nivolumab
All-Cause Mortality (participants affected / at risk) | 14/17 | 3/8
Serious Adverse Events (participants affected / at risk) | 3/17 | 5/8
Other Adverse Events (participants affected / at risk) | 17/17 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: RXC004 Monotherapy (N=17) | Arm B: RXC004+Nivolumab (N=8)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: RXC004 Monotherapy (N=17) | Arm B: RXC004+Nivolumab (N=8)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (15) | 4 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 5 (7)
Vomiting (Gastrointestinal disorders) | 4 (10) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 4 (5)
Asthenia (General disorders) | 4 (4) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Stoma prolapse (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (3) | 4 (4)
Blood bilirubin increased (Investigations) | 2 (2) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Amylase increased (Investigations) | 2 (2) | 0 (0)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (2)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (1)
Carcinoembryonic antigen increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Gastric pH decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Urine calcium decreased (Investigations) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 5 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 9 (11) | 6 (7)
Lethargy (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT04907539/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT04907539/SAP_001.pdf